CLINICAL TRIAL: NCT01384006
Title: EXTENDED PANCREAS DONOR PROGRAM - THE EXPAND STUDY
Acronym: EXPAND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Collaborators: Charite University, Berlin, Germany (Other); Ludwig-Maximilians - University of Munich (Other); University of Jena (Other); Johann Wolfgang Goethe University Hospital (Other); University Hospital Tuebingen (Other); University Hospital Erlangen (Other); University of Heidelberg Medical Center (Other); University of Leipzig (Other); University Hospital Dresden (Other); University Hospital Bergmannsheil Bochum (Other); Hannover Medical School (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University of Kiel (Other); Transplantationszentrum Köln-Merheim (Other)
Responsible Party: Regensburg University Hospital, UKR
Other Study IDs: EXPAND
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Pancreas Allograft Recipients w/wo Kidney Transplantation
Keywords: Pancreas transplantation; extended donor criteria; organ survival

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: standard pancreas allograft recipients
- Study: recipients of extended donor criteria pancreas allografts

SUMMARY:
To expand the donor pool for pancreas allografts. For detailed description please see below.

DETAILED DESCRIPTION:
This is an investigator initiated prospective, non-randomized feasibility-study, comparing recipients of EDC-pancreas allografts (SPK or PTA) with patients undergoing SPK or PTA with standard criteria allografts.

Simultaneous Pancreas Kidney transplantation (SPK) or Pancreas Transplantation alone (PTA) are life saving procedures for patients with type 1 (juvenile) diabetes mellitus and impaired renal function. Although the waiting lists for SPK and PTA are increasing, the numbers of pancreas transplantations are declining in the Eurotransplant (ET) area (www.eurotransplant.nl). One major reason for this decline is the fact that a large number of pancreas allografts, potentially eligible for transplantation are excluded by the ET pancreas allocation system (EPAS). Those criteria include an organ-specific cut-off for donor age >50 years and/or BMI>30. This means that donors that are older than 50 years or donors with a BMI >30 are, at the moment, not considered for solid organ transplantation. The pancreas will be directly allocated for islet transplantation (Eurotransplant manual - version may 26, 2009).

The organ-specific cut-off was once established to provide donor pancreases for islet transplantation. Although 173 pancreases were allocated and retrieved for islet transplantation only 17 islet transplantations were performed in the whole ET area in 2008 (ET data). In Germany two islet transplantations were performed in 2009. Best results after islet transplantation are achieved with organs obtained from young obese donors. Concerning allocation, no conflict of interest exists between whole organ and islet transplantation, the single active German islet center will take part in the EXPAND study. Meanwhile, according to the suggestions by the EXPAND study group, extended donor pancreases are intended to be offered regionally as "rescue" allocation to the centers. The centers should then decide if this organ can be transplanted as whole organ or if it can be used for islets.

As the average age for a post mortal organ donor in the ET area is now 58 years, there is a severe donor selection by age leading to organ shortage. In Germany in 2008 the total number of organ donors was 1.198. However, only 510 donors had an age between 3 and 50 years and thus were potentially eligible for pancreas donation. Out of the 510 donors only 183 pancreases (36% of all potential, age restricted pancreas donors) were retrieved and 127 (25%) were transplanted (DSO, Deutsche Stiftung für Organtransplantation e.V.). Altogether, 676 donors were not even screened for pancreas donation due to age, regardless to all other medical conditions. In addition, approximately 13% were not eligible for pancreas donation only due to BMI. Moreover, in the ET-area pancreases are allocated without local priority leading to longer ischemic times due to transport ways. However, there are data from other allocation areas throughout the world (UNOS or UK) showing that a good overall outcome after PTx can be achieved with donors exceeding the defined allocation criteria defined by ET (older than 50 or BMI>30), if the cold ischemic time is kept short. In Great Britain, a local retrieval and allocation system was installed in 2000 resulting in a steep increase in pancreas transplantation. Moreover, within this new allocation system the currently worldwide largest and most successful pancreas transplant program was initiated in Oxford in 2004 with an extensive use of extended pancreas donors leading to excellent results. These extended criteria avoided donor BMI restriction, and accepted donors with an age between 8 and 68 years. Meanwhile 350 SPK and PTA were transplanted with an excellent one year pancreas survival of 91%, kidney survival 95% and a patient survival of 96%.

In the US, a retrospective analysis of OPTN registries compared 8.850 SPK from young donors vs. 776 SPK from donors >45 years. It showed that patients transplanted from an older donor have equal survival compared to those who were waiting for a young donor for more than 1.5 years. However the earlier transplanted patient is instantly off dialysis and insulin. Good results were already achieved with extended pancreas donors in the US and also in one German study.

Based on those findings, a new pancreas allocation system was established in the USA where standard pancreases (donor age < 50y or BMI < 30) are allocated first on local, then on regional and then on national levels and extended pancreas (donor age > 50 years or BMI > 30) are allocated locally only.

In conclusion, these data indicate the requirement for a new allocation system also in the ET area to be able to provide a sufficient number of organs for patients on the waiting list. We therefore suggest a new pancreas allocation system where donors with an age of 50-60 years or a BMI of 30-34 are allocated regionally within a cold ischemic time < 12 h. To prove the hypothesis that extended pancreas allograft donors can be used safely with equal outcome in recipients a prospective comparative multicenter feasibility-study is required.

A good example of a successful change of allocation rules is the European Senior Donor Program (ESDP) for kidneys, the so called "old for old" program. Within this program kidneys from donors >65 years are allocated regionally to patients >65 years with a relatively short ischemic time without HLA matching. For this purpose a comparative study was performed to prove the efficacy of this allocation change.

The standard immunosuppression for SPK or PTA includes induction therapy with antibodies. Maintenance therapy is mostly performed with a tacrolimus / mycophenolate mofetil combination. The usage of calcineurin inhibitors for maintenance therapy is characterized by a clear transition from cyclosporine to tacrolimus. Myfortic® vs. Cell Cept® shows beneficial effects after SPK in a large single center comparison. Corticosteroids are administered to the majority of patients; however, steroid-avoidance and steroid-withdrawal protocols are increasingly common.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of standard allocation organs or
* Recipients of organs from donors between 50 to 60 years OR a BMI 30-34
* CIT (cold ischemic time) ≤ 12h (only local allocation of organs, optimally the procuring surgical team should be the transplanting team).

and

* negative cross-match
* age > 18 years
* primary SPK, PAK or PTA
* Patients on standardized immunosuppressive treatment with Tacrolimus (Prograf®), MPA (Myfortic®) [aiming at center specific trough-level practice] from day 5 after transplantation (prior to day 5 MMF (Cell Cept®) can be applied as i.v. medication due to reduced gastrointestinal passage and insecure absorption of orally applied medication) and center-specific steroid treatment.

Exclusion Criteria:

* Malignant diseases within 5 years prior to PTA/SPK except for squamous cell carcinoma and basalioma of the skin.
* Pancreas retransplantation.
* Immunized patients with a preformed antibody titer>5%.
* Women with child bearing potential.
* Patients with a psychological, familial, sociologic or geographic condition potentially hampering compliance with the study protocol and follow-up schedule.
* Patients under guardianship (e.g. individuals who are not able to freely give their informed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreas allograft recipients in Germany
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Pancreas allograft survival at 3 months after transplantation | 3 months
  Pancreas allograft survival at 3 months after transplantation has been defined as primary endpoint. Patients that are insulin-free and have a normal fasting glucose level 60 - 140 mg/dl (3.3 - 7.8 mmol/l) in peripheral venous blood are regarded as having a functioning organ. Thus, all patients that have a pathologic fasting glucose level at 3 months will be counted as event with regards to the primary endpoint of pancreas allograft survival.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan A Farkas, MD, Study Director — Regensburg Univeristy Hospital; Andreas A Schnitzbauer, MD, Principal Investigator — Regensburg University Hospital
Locations (1):
- Regensburg University Hospital, Regensburg, Bavaria, Germany

REFERENCES:
- [Derived] Proneth A, Schnitzbauer AA, Schenker P, Wunsch A, Rauchfuss F, Arbogast H, Manekeller S, Nadalin S, Heise M, Strohlein MA, Banas B, Schemmer P, Becker T, Bechstein WO, Pascher A, Viebahn R, Geissler EK, Schlitt HJ, Farkas SA. Extended Pancreas Donor Program-The EXPAND Study: A Prospective Multicenter Trial Testing the Use of Pancreas Donors Older Than 50 Years. Transplantation. 2018 Aug;102(8):1330-1337. doi: 10.1097/TP.0000000000002122. PMID 29406443
- [Derived] Proneth A, Schnitzbauer AA, Zeman F, Foerster JR, Holub I, Arbogast H, Bechstein WO, Becker T, Dietz C, Guba M, Heise M, Jonas S, Kersting S, Klempnauer J, Manekeller S, Muller V, Nadalin S, Nashan B, Pascher A, Rauchfuss F, Strohlein MA, Schemmer P, Schenker P, Thorban S, Vogel T, Rahmel AO, Viebahn R, Banas B, Geissler EK, Schlitt HJ, Farkas SA. Extended pancreas donor program - the EXPAND study rationale and study protocol. Transplant Res. 2013 Jul 1;2(1):12. doi: 10.1186/2047-1440-2-12. PMID 23816330